CLINICAL TRIAL: NCT04067232
Title: 4 Dimensional - Impairment of Posttraumatic Forearm Rotation Evaluated With Computed Tomography : 4D-IRECT Pilot Trial
Brief Title: 4 Dimensional - Impairment of Posttraumatic Forearm Rotation Evaluated With Computed Tomography
Acronym: 4D-IRECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL18_0463; UF 7729 (Other: Sponsor)
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2020-09

CONDITIONS: Pronation-Supination of the Forearm, Impairment of
Keywords: Four Dimensional Computed Tomography (4D-CT)
MeSH Terms: conditions — Pronation-Supination Of The Forearm, Impairment Of | interventions — Four-Dimensional Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with posttraumatic forearm impairment (Experimental): All patients with a one-sided posttraumatic impairment of forearm pro- and/or supination at least 3 months after injury
  Interventions: Diagnostic Test: 4D-CT-scan

INTERVENTIONS:
Diagnostic Test: 4D-CT-scan — Both forearms of the subjects with posttraumatic forearm impairment are scanned with a 4D-CT scanning technique, during forearm rotation.

SUMMARY:
The aim of this study is to develop a 4D-CT (4 Dimensional Computed Tomography) -scan acquisition method for estimating the cause of posttraumatic impairment of the forearm. Both forearms of patients with posttraumatic impairment of one of the forearm will be scanned using a 4D-CT-scan, during forearm rotation. Rotation of impaired and healthy forearms will be analysed and compared to each other. This method is intended to allow differentiation of motion patterns reflecting an osseous impairment from those caused by soft tissue pathology in order to improve treatment choice.

DETAILED DESCRIPTION:
Forearm and wrist fractures are the most common of all fractures and mostly occur at the distal end of the radius. Distal radius fractures are associated with posttraumatic sequelae, which typically involve restricted forearm rotation. Diagnostics of dynamic traumatic pathologies are conventionally based on static (2D or 3D) imaging protocols using MRI (magnetic resonance imaging) or CT. However, interpretation of indirect suggestive findings - such as edema or abnormal bone positions - limits accuracy and inter-observer reliability. Dynamic 4D imaging (adding the fourth dimension of time) has the potential to discriminate whether forearm rotation deficit is due to an osseous deformity causing bony impingement or whether it is due to non-osseous pathology. Hence it may reduce unnecessary corrective osteotomies and guide the patient and surgeon towards the most effective surgical or conservative treatment choice - expectedly resulting in better outcomes and patient satisfaction. In addition, we aim to develop a classification based on the estimated motion patterns and assess its reliability. Furthermore we aim at acquiring knowledge of physiological mechanics of the radioulnar joint and to assess symmetry in radioulnar joint motions between two healthy forearms on 4D-CT-scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a one-sided posttraumatic impairment of forearm pro- and/or supination at least 3 months after injury
* Patients are above 18 years
* Patients who are willing to give informed consent
* National health insurance cover

Exclusion Criteria:

* A history of trauma to both forearms
* Any shoulder pathology or impairment preventing forward elevation of the arm as required during the scanning protocol
* Neuromuscular pathology
* Not able to understand or give informed consent
* Pregnancy (βHCG positive), breast-feeding or the absence of effective contraception for women of child-bearing age
* Legal incapacity (persons in custody or under guardianship)
* Deprived of liberty Subject (by judicial or administrative decision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Quantification of forearm motion patterns | the 4D-CT-scan procedure
  Calculate the mean and standard deviation of the healthy versus the affected forearm rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Geert BUIJZE, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No